CLINICAL TRIAL: NCT05276817
Title: Microbiological Evaluation of Diode Laser Bacterial Reduction as Adjunct to Periodontal Maintenance Treatment: A Pilot Clinical Study
Brief Title: Perio. Maint. With Diode LBR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biolase Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOL-LBR-P-2022
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: Split mouth study. For each patient, each quadrant is assigned to a randomized treatment. 4 treatment arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Perio maint. then sham laser (Sham Comparator)
  Interventions: Device: Sham
- Perio maint. then medicament (Experimental)
  Interventions: Drug: HP
- Perio maint. then diode laser 1 (Experimental)
  Interventions: Device: Epic Diode
- Perio maint. then diode laser 2 (Experimental)
  Interventions: Device: Epic Diode

INTERVENTIONS:
Device: Epic Diode — HP solution will be inserted to the bottom of the periodontal pocket using a disposable side port needle applicator. The diode tip will be inserted into the pocket, parallel with the root surface and moved in slow side to side motions, painting in the full depth and width of the pocket while activating the diode laser.
  Arms: Perio maint. then diode laser 1; Perio maint. then diode laser 2
Drug: HP — HP solution will be inserted to the bottom of the periodontal pocket using a disposable side port needle applicator. The solution will be in the pocket for 30 seconds, and then removed using sterile gauze and water spray.
  Arms: Perio maint. then medicament
Device: Sham — The diode tip will be inserted into the pocket, parallel with the root surface and moved in slow side to side motions, painting in the full depth and width of the pocket. The diode laser will not be activated during the sham treatment. Coe-Pak periodontal dressing will be applied to the control quadrant to isolate it.
  Arms: Perio maint. then sham laser

SUMMARY:
The primary aim of this pilot study is to determine whether the test methods described feasibly achieve the goal defined for a future clinical study. The purpose is a quantitative assessment of the bactericidal effect of two adjunctive treatments compared to that of conventional periodontal maintenance debridement. Patients who meet eligibility criteria and are enrolled in the study will receive the standard of care, whole mouth periodontal maintenance treatment using ultrasonic scalers to debride deposits within the gingival sulcus. Subsequently, each of three of the quadrants will be randomly assigned to a test group (keeping the fourth quadrant as the control), thus, a "split-mouth" study design. Microbial samples will be collected using sterile paper points inserted into each tooth site involved in the study at baseline (S1) before test treatment and one week after test treatment (S2). Samples will be analyzed with real time qPCR to identify and quantify specific periodontal pathogens. Data analysis will compare the post-treatment results to baseline, the control treatment arm to the test treatment arm, and the test treatments among each other.

ELIGIBILITY:
Inclusion Criteria:

* • Adults, over 30 years old

  * At least one site in each quadrant having CAL 4-6mm and/or PPD 5-7mm (at least 4 sites per patient) with all adjacent sites having PPD<5mm
  * Patients who received SRP treatment in the past 12 months, who are returning for routine periodontal maintenance debridement, whose pockets are stable at PPD 5-7mm (not showing improvement or decline)

Exclusion Criteria:

* • Patients who have had periodontal surgery within 12 months

  * A site adjacent to the potential study site having either an implant placed or a PPD>7mm
  * Patients taking systemic antibiotics or immunosuppressants during or within 3 months of the study
  * Chronic smokers or smokeless tobacco users

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Bacteria concentration measured by qPCR | 1 week
  Change in levels of the total bacterial load and of individual bacteria from baseline and compared to control.

SECONDARY OUTCOMES:
Incidence of adverse events | 3 months
  Monitoring of patient acceptance of the adjunctive treatment and monitoring of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Stephen John, DDS, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No